CLINICAL TRIAL: NCT06896045
Title: Multicenter Study Evaluating the Relationship Between Perceived Daily Stress Level and Glycemic Level in Subjects With Type 1 Diabetes
Acronym: EVASTRESS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre d'Etudes et de Recherche pour l'Intensification du Traitement du Diabète (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2024-A02296-41
Record Dates: First submitted 2025-02-28; First posted 2025-03-26 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Diabetes Type 1
Keywords: stress; glycemic control
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Visual analog scale to measure stress levels (Experimental)
  Interventions: Behavioral: Assess stress levels 4 times a day before meals (morning, noon and evening and at bedtime) using a visual analogue scale

INTERVENTIONS:
Behavioral: Assess stress levels 4 times a day before meals (morning, noon and evening and at bedtime) using a visual analogue scale — In addition to stress assessment with the stress meter, patients will be fitted with a Continious Glucose Monitoring

SUMMARY:
Type 1 diabetes (T1D) affects around 200,000 people in France. The only treatment is insulin, administered either by multiple injections, by pump alone or, more recently, by automated insulin delivery systems (AIDs), which have resulted in a very significant improvement in glycaemic control and quality of life. These closed-loop (CL) devices are capable of effectively regulating the conventional factors associated with glycaemic disturbance, namely dietary intake and physical activity. However, they do not account of stress, which some subjects with T1D perceive as a major disrupter of their blood sugar levels. One of the reasons for this is undoubtedly that stress, unlike diet or physical activity, cannot be anticipated. Since stress is difficult to predict, it is also more difficult to study. Its onset, intensity, duration and progression are linked to the subject's experience, psychological state and environment. Not all patients respond to stress triggers in the same way. Some patients appear to be more reactive than others to these agents, particularly when they are exposed to them chronically or repeatedly, in an anxiety-provoking environment. This is known as chronic psychosocial stress, and it is this type of stress that seems to be most closely associated with glycaemic disturbance in subjects with T1D, most often in the form of hyperglycaemia and, more rarely, hypoglycaemia. However, there are no solid epidemiological or experimental data to support these observations.

The study we propose is a prospective multicentre clinical trial in 125 subjects with T1D treated with insulin pumps or multi-injections at 14 French university centres. Our aim is to evaluate the relationship between interstitial glucose levels measured by CGM and perceived stress, assessed 4 times a day, away from mealtimes in order to avoid the impact of dietary glycaemia, using a "stressometer". This stressometer is an application designed by CERITD that can be downloaded to the patient's smartphone and consists of an electronic visual analogue scale (VAS) on which the level of stress felt is evaluated quantitatively (continuous value between 0 and 10).

ELIGIBILITY:
Inclusion Criteria:

* Patient with a clinical diagnosis of type 1 diabetes of at least 1 year, as determined by the medical record;
* Patient aged at least 18 years;
* Patient treated with an external insulin pump for at least 2 months or with multi-injections;
* Patient with a smartphone compatible with iOS 15.0 or higher or Android 12.0 or higher;
* Patient with a smartphone with Bluetooth 5.0 or higher;
* Patient with HbA1c ≤ 10% with measurement ≤3 months;
* Patient with no psychiatric pathology that could interfere with the study;
* Patient having signed the free and informed consent form to participate in the study;
* Patient affiliated to the French Social Security system;
* Patient agreeing not to eat between meals for the duration of the study (except for hypoglycaemia and/or snacks during physical activity);
* Patient agrees to wear an Empatica EmbracePlus watch for the duration of the study and to charge it according to the device's requirements for recording data;
* Patient agreed to wear an OURA ring for the duration of the study and to recharge it as required by the device to enable data recording (patients at the CERITD centre only).

Exclusion Criteria:

* Type 2 diabetic patient;
* Patient fitted with a closed loop (or artificial pancreas);
* Patient with any characteristic pathology that could interfere with the study (renal failure, unstabilised diabetic retinopathy, heart failure, heart attack within 6 months prior to inclusion, severe neuropathy, particularly autonomic neuropathy);
* Patients with a tendency to snack;
* Patients undergoing treatment with drugs known to significantly interfere with blood sugar levels or the adrenergic system, such as corticosteroids and beta-blockers;
* Patients undergoing atropine treatment (Hydroxyzine Chlorhydrate or Atarax®...), likely to modify the EDA (Electrodermal Activity) ;
* Patients with a known allergy to latex (watch EmbracePlus);
* Pregnant woman;
* Nursing woman;
* Persons deprived of their liberty by judicial or administrative decision, persons under psychiatric care;
* Persons under guardianship or trusteeship or subject to a legal protection measure
* Persons who are not affiliated to a social security scheme or are beneficiaries of such a scheme.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2025-04-22 (Actual); Primary Completion 2026-02-05 (Estimated); Study Completion 2026-02-05 (Estimated)

PRIMARY OUTCOMES:
Correlation between perceived daily stress, self-assessed on a multi-daily basis using a mobile subjective stress assessment application called a "stress meter", and blood glucose levels measured by continuous glucose monitoring (CGM) | 14 days
  Visual analogue scale to assess stress levels:
  0: I feel absolutely no stress 10: I feel extremely stressed

SECONDARY OUTCOMES:
HbA1c measurement | At Inclusion
  HbA1c measurement at inclusion
Characterization of 4 patient profiles according to the impact of daily stress on glycemic control | At inclusion
  Questionnaire for Assessing the Impact of Stress on Blood Sugar Levels. This questionnaire was designed and developed by CERITD to assess the impact of perceived stress on blood glucose levels in T1DM patients.
Number of days the Continuous subcutaneous Glucose Monitoring (CGM) worn | 14 days
Percentage of time the CGM is active (recommended at least 70% of the time) | 14 days
Percentage of sensor time in glucose level measured by the Dexcom One+ CGM time | 14 days
  * Percentage of time spent within the target 70-180 mg/dl (3.9-10.0 mmol/L) (TIR)
  * Percentage of time <54 mg/dl (<3.0 mmol/L)
  * Percentage of time spent in the range 54-69 mg/dl (3.0-3.8 mmol/L)
  * Percentage <70 mg/dl (<3.9 mmol/L)
  * Percentage of time >250 mg/dl (>13.9 mmol/L)
  * Percentage of time spent in the range 181-250 mg/dl (10.1-13.9 mmol/L)
  * Percentage of time >180 mg/dl (>10.0 mmol/L)
Variability of the CGM glucose level | 14 days
  The glycemic variation coefficient (CV) intra patient CV≤36%, CV > 36%
Glucose management Indicator (GMI) | 14 days
Average CGM glucose level | 14 days
  Measurement of glucose by CGM
Glycaemic evolution over a period during which stress is measured. | 14 days
  Measurement of the area under the curve (AUC) for blood glucose
Glycaemic evolution over a period during which stress is measured. | 14 days
  Measurement of the maximum blood sugar
Glycaemic evolution over a period during which stress is measured. | 14 days
  Measurement of the blood sugar delta
Glycaemic evolution over a period during which stress is measured. | 14 days
  Measurement of the blood sugar average
Measuring heart rate with the Empatica EmbracePlus watch | 14 days
Measuring heart rate variability with the Empatica EmbracePlus watch | 14 days
Measuring electrodermal activity with the Empatica EmbracePlus watch | 14 days
Measuring heart rate with the Oura ring | 14 days
Measuring heart rate variability with the Oura ring | 14 days
Measuring accelerometry parameters with the Empatica EmbracePlus watch | 14 days
Measuring accelerometry parameters with the Oura ring | 14 days
Measuring the amount of sleep you get with the Empatica EmbracePlus watch | 14 days
  "Sleep detection" parameter
Measuring the amount of sleep you get with the Oura ring | 14 days
  sleep score
Measuring total sleep time with the Oura ring | 14 days
Assessment of sleep quality | 14 days
  Visual Analogue Sleep Scale filled in each morning with reference to the previous night 0: I slept very badly 10: I slept very well
Measurement of sleep characteristics with the Oura ring | 14 days
  Sleep efficiency as a percentage
Measurement of inflammatory biomarkers | at inclusion and after 14 days
Capillary cortisol measurement | After 14 days
  Hair cortisol levels measured at the end of study.
Assessment of diabetes-related distress in the test population . | at inclusion
  PAID (Problem Areas in Diabetes) is a self-administered 5-item scale. Each item is scored from 0 (not a problem) to 4 (serious problem).
Assessment of stress levels using the STAI questionnaire | At inclusion and after 14 days
  State-Trait Anxiety Inventory (STAI)-Y1:
  The STAI-Y1 is composed of 20 items. This questionnaire assesses how the patient feels at the present moment. Patients are asked to score each question on a four-point scale (from 1 -corresponding to "not at all" to 4 - "much").
Assessment of stress levels using the STAI questionnaire | After 14 days
  State-Trait Anxiety Inventory STAI-Y2 (anxiety score): The STAI-Y2 is composed of 20 items. This questionnaire assesses how the patient feels in general. Patients are asked to answer each question on a four-point scale (from 1 - corresponding to "almost never" to 4 -"almost always")
Assessment of diabetes-related distress in the test population . | at inclusion and after 14 days
  DDS T1 is an indicator of overall diabetes distress (average of 17 items, rated 1 to 6 on a scale).
  A higher score indicates higher distress.
Evaluation of the perception of hypoglycaemia in the population tested with Clarke score | at inclusion
  The Clarke questionnaire is comprised of eight questions to evaluate the hypoglycemia awareness. The answer for each individual question will represent a score (0 or 1). These scores will be summed together to a final score from 0 to 7, representing from normal to minimal/no hypoglycemia awareness.
Evaluation of the perception of hypoglycaemia in the population tested with Gold score | at inclusion
  The Gold method is used to assess impaired awareness of hypoglycemia. The scale is from 1 to 7. A score of 4 or more indicates impaired awareness of hypoglycemia
Assessment of stress levels using the PSS-14 questionnaire (Perceived Stress Scale 14) | at inclusion and after 14 days
  It is a five-point Likert-type scale and consists of 14 items. Participants rate each item on a scale ranging from "Never (0)" to "Very often (4)". Seven of the items with positive statements are scored in reverse. As the scores obtained from the scale increase, the perceived stress level of the person increases. PSS-14 scores range from 0 to 56, with 0-35 point range indicating normal stress level, 35-56 point range indicating that the individual is under stress
Assessment of stress levels : depression score | After 7 days
  The Depression, Anxiety and Stress Scale 21 (DASS-21) is an inventory that will be used to identify the presence and intensity of depressive, anxiety and stress. For depression the cutoff scores are: Normal: 0-9, Mild: 10-12, Moderate:13-20, Severe: 21-27, and Extremely severe: 28-42.
Assessment of stress levels : anxiety score | After 7 days
  The Depression, Anxiety and Stress Scale 21 (DASS-21) is an inventory that will be used to identify the presence and intensity of depressive, anxiety and stress. For anxiety the cutoff scores are: Normal: 0-6, Mild: 7-9, Moderate: 10-14, Severe:15-19, and Extremely severe: 20-42.
Assessment of stress levels : stress score | After 7 days
  The Depression, Anxiety and Stress Scale 21 (DASS-21) is an inventory that will be used to identify the presence and intensity of depressive, anxiety and stress. For stress the cutoff scores are: Normal: 0-10, Mild:11-18, Moderate:19-26, Severe: 27-34, and Extremely severe: 35-42.
Diagnosis and measurement of the severity of depression: Patient Health Questionnaire (PHQ-9) | After 7 days
  The Patient Health Questionnaire (PHQ-9) will be used to assess depressive symptoms, including suicidal ideation, over the last two weeks (9 questions). Items are scored 0-3, resulting in a total score of 0-27. Higher scores indicate more symptoms of depression.
Personality traits : Big Five Inventory 10 (BFI-10) | After 7 days
  Items range from 1 (strongly approves) to 5 (strongly disapproves). Scales: openness to experience, conscientiousness, extraversion, agreeableness and neuroticism
Bortner scale | After 7 days
  The Bortner self-assessment questionnaire consists of 14 items. It is used to classify individuals according to types of behaviour (A and B)
Quality of life assessment: Short Form 36 questionnaire (SF-36) | After 14 days
  Short Form 36 (SF-36) -ranges between 0 (maximum disability) and 100 (no disability). The SF36 score can be converted to utility scores using values within the questionnaire.
Assessment of sleep quality: Pittsburgh Sleep Quality Index (PSQI) | After 14 days
  Pittsburgh Sleep Quality Index (PSQI), a self-report questionnaire comprising seven component scores (subjective sleep quality, sleep latency, duration of sleep, sleep efficiency habits, sleep disturbances, use of sleeping medication, and daytime dysfunction), is used to evaluate sleep quality over the last month

CONTACTS AND LOCATIONS:
Overall Officials: Sylvia Franc, MD, Principal Investigator — Centre d'Etudes et de Recherche pour l'Intensification du Traitement du Diabète
Locations (14):
- France (14):
  - Angers University Hospital, Angers
  - Avignon Hospital, Avignon
  - Bordeaux University Hospital, Bordeaux
  - Brest University Hospital, Brest
  - Dijon University Hospital, Dijon
  - CERITD (Centre d'Etudes et de Recherches pour l'Intensification du Traitement du Diabète), Évry
  - Grenoble University Hospital, Grenoble
  - St Louis Hospital, La Rochelle
  - Lille University Hospital, Lille
  - DiabeCare diabetes centre, Lyon
  - European Hospital, Marseille
  - Private practice in endocrinology and metabolic diseases, Mérignac
  - Rennes University Hospital, Rennes
  - Strasbourg University Hospital, Strasbourg

IPD SHARING:
Plan to Share IPD: No